CLINICAL TRIAL: NCT00455741
Title: Effect of Age on Gonadotropin Responses to Short-Term Negative and Positive Feedback Effects of Gonadal Steroids Using PET Scanning
Brief Title: Postmenopausal Women Estrogen and Progesterone Infusion
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Janet E. Hall, MD, Associate Physician, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2000P-002496; R01AG013241 (NIH)
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Results first posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-04

CONDITIONS: Postmenopause; Aging
Keywords: menopause; estrogen; progesterone; hormone replacement; aging; PET

STUDY DESIGN:
Intervention Model Description: Estradiol and progesterone infusion to assess negative and positive feedback on the hypothalamus and pituitary in young and older postmenopausal women.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Young postmenopausal women (Active Comparator): Graded estradiol infusion to young postmenopausal women. Graded progesterone infusion to young postmenopausal women.
  Interventions: Drug: Estradiol infusion; Drug: Progesterone infusion
- Older postmenopausal women (Active Comparator): Graded estradiol infusion to young postmenopausal women. Graded progesterone infusion to young postmenopausal women..
  Interventions: Drug: Estradiol infusion; Drug: Progesterone infusion

INTERVENTIONS:
Drug: Estradiol infusion — Graded estradiol infusion of 0.1 mcg/kg/hr for 12 hr, 0.135 mcg/kg/hr for 12 hr, 0.165 mcg/kg/hr for 12 hr and 0.2 mcg/kg/hr for 60 hr.
Drug: Progesterone infusion — Progesterone infusion of 4.77 nmol/kg/hr (1.5 mcg/kg/hr) for 24 hr and 6.36 nmol/kg/hr (2 mcg/kg/hr) for the final 24 hr of the 5-day study.

SUMMARY:
The purpose of the study is to study the effects of aging, estrogen and progesterone on the brain. Specifically, we want to look at how the hypothalamus and pituitary (two small glands in the brain) respond to estrogen. The pituitary gland is controlled by the hypothalamus. The hypothalamus secretes GnRH (Gonadotropin-Releasing Hormone) that signals the pituitary to secrete the reproductive hormones, LH (Luteinizing Hormone) and FSH (Follicle Stimulating Hormone). These hormones act on the ovaries and signal the ovaries to produce estrogen and progesterone. Estrogen in the bloodstream then acts on the brain to modulate this system with changes in LH and FSH. Early changes associated with low levels of estrogen are inhibitory (estrogen negative feedback) while higher levels of estrogen (such as those present when a follicle in the ovary is ready to ovulate) stimulate LH to cause ovulation (positive feedback). This study will determine: 1) hypothalamic and pituitary levels of glucose uptake (as a measure of brain metabolic activity) at baseline and in association with estrogen negative feedback on LH (24 hr) and estrogen positive feedback on LH (72 hr); and 2) the effect of aging on estrogen feedback on LH, assessing negative feedback (nadir ~ 24 hr) and positive feedback (peak between 72 and 96 hr).

DETAILED DESCRIPTION:
The transition to menopause is characterized by a decline in the numbers of functional ovarian follicles followed by a decrease in levels of inhibin A and B and complex changes in estradiol, which include an initial increase followed by an inevitable decrease. Therefore, there are dynamic changes in the hypothalamic-pituitary feedback from the aging ovary, prior to the ultimate loss of feedback that occurs with the complete cessation of ovarian function. While there is ample evidence that the loss of ovarian function is a major contributor to the menopause, there is evidence from animal models that primary age-related neuroendocrine changes may also contribute to reproductive aging. Specifically, there is evidence for changes in the hypothalamic and pituitary responses to estrogen negative and positive feedback. An understanding of the age-related changes in the physiology of the hypothalamic and pituitary responsiveness to gonadal steroid feedback is critical in determining whether hypothalamic and pituitary changes per se contribute to the menopause and the impact of the loss of reproductive function on the brain.

ELIGIBILITY:
Inclusion criteria:

postmenopausal women young (age 45-55) or old (age 70-80) History of natural menopause defined by the absence of menses for at least 12 months (or history of surgical menopause defined as bilateral oophorectomy) Normal TSH, PRL and CBC, and Factor V activity Normal BUN and Creatinine (< 2 times the upper limit of normal) BMI between 18 to 30 kg/m2 An increased FSH measured at the screening visit will be consistent with menopause. If the initial determination is low, a repeat sample may be drawn.

Exclusion criteria:

Hormonal medication or herbal supplements and/or over the counter menopause therapy in the 2 months prior to study Any absolute contraindications to the use of physiologic replacement doses of estrogen and/or progesterone History of coronary artery disease Medications thought to act centrally on the GnRH pulse generator History of breast cancer or blood clots Smoking more than 10 cigarettes/day Prior history of allergic reaction to any dyes used with x-rays or scans and/ or any other contraindications to PET scans No metal implants, pacemakers, aneurysm clips, implanted hearing aids and/or any other contraindications to MRI scan

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2000-11; Primary Completion 2007-02 (Actual); Study Completion 2015-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet E Hall, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Requests for sharing coded results without patient identifiers can be made directly to the PI.

REFERENCES:
- [Result] Shaw ND, Srouji SS, Histed SN, Hall JE. Differential effects of aging on estrogen negative and positive feedback. Am J Physiol Endocrinol Metab. 2011 Aug;301(2):E351-5. doi: 10.1152/ajpendo.00150.2011. Epub 2011 May 10. PMID 21558550
- [Result] Ottowitz WE, Derro D, Dougherty DD, Lindquist MA, Fischman AJ, Hall JE. FDG-PET analysis of amygdalar-cortical network covariance during pre- versus post-menopausal estrogen levels: potential relevance to resting state networks, mood, and cognition. Neuro Endocrinol Lett. 2008 Aug;29(4):467-74. PMID 18766152
- [Result] Ottowitz WE, Dougherty DD, Fischman AJ, Hall JE. [18F]2-fluoro-2-deoxy-D-glucose positron emission tomography demonstration of estrogen negative and positive feedback on luteinizing hormone secretion in women. J Clin Endocrinol Metab. 2008 Aug;93(8):3208-14. doi: 10.1210/jc.2008-0203. Epub 2008 Jun 3. PMID 18522979
- [Result] Ottowitz WE, Siedlecki KL, Lindquist MA, Dougherty DD, Fischman AJ, Hall JE. Evaluation of prefrontal-hippocampal effective connectivity following 24 hours of estrogen infusion: an FDG-PET study. Psychoneuroendocrinology. 2008 Nov;33(10):1419-25. doi: 10.1016/j.psyneuen.2008.09.013. Epub 2008 Oct 31. PMID 18977091

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 36 subjects consented; 6 failed screening, 2 decided not to participate.
Pre-assignment Details: 1 subject terminated during study (hemoglobin drop) for a total of 24 completed.
Groups:
- Younger PMW: Postmenopausal women (PMW) ages 45-55 receiving the following hormone infusions.
  Estradiol infusion:
  Graded estradiol infusion of 0.1 mcg/kg/hr for 12 hr, 0.135 mcg/kg/hr for 12 hr, 0.165 mcg/kg/hr for 12 hr, and 0.2 mcg/kg/hr for 60 hr.
  Progesterone infusion:
  Progesterone infusion of 4.77 nmol/kg/hr (1.5 mcg/kg/hr) for 24 hr and 6.36 nmol/kg/hr (2 mcg/kg/hr) for the final 24 hr of the 5-day study.
- Older PMW: Postmenopausal women (PMW) ages 70-80 receiving the following hormone infusions.
  Estradiol infusion:
  Graded estradiol infusion of 0.1 mcg/kg/hr for 12 hr, 0.135 mcg/kg/hr for 12 hr, 0.165 mcg/kg/hr for 12 hr, and 0.2 mcg/kg/hr for 60 hr.
  Progesterone infusion:
  Progesterone infusion of 4.77 nmol/kg/hr (1.5 mcg/kg/hr) for 24 hr and 6.36 nmol/kg/hr (2 mcg/kg/hr) for the final 24 hr of the 5-day study.
Period: Overall Study
Arm/Group | Younger PMW | Older PMW
Started | 13 | 12
Completed | 13 | 11
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects were healthy and had experienced their last menstrual period 18 mo previously. Subjects were not on any medications known to interact with the neuroendocrine reproductive axis, including over-the-counter medications or herbal remedies. Factor V Leiden mutations were absent in all patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Younger PMW | Older PMW | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Customized [Mean (Standard Deviation); unit: years] | 49.9 (3.8) | 75.2 (3.6) | 61.3 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 0 | 5
  White | 8 | 12 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 20

OUTCOME MEASURES:

1. Primary Outcome: Effect of Aging on Estrogen Negative Feedback on LH
Description: Difference between baseline LH (average of 3 samples drawn 15 min apart) and nadir LH based on a 3-point moving average of blood samples drawn every 4 hours over 120 hr, expressed as a percent of baseline (% baseline).
Time Frame: Baseline at 0 time before infusion, nadir occurred between 8 and 60 hr (mean 24 hr)
Population: NOTE: 2 older and 2 younger postmenopausal women excluded from this analysis as estradiol levels exceeded physiological exposure levels
Measure: Mean (Standard Error); unit: % change from baseline
Arm/Group | Younger PMW | Older PMW
Number analyzed (Participants) | 11 | 9
% change from baseline | -52.8 (3.0) | -53.2 (2.3)
Statistical Analysis 1: Comparison: Younger PMW vs Older PMW; effect of age on estrogen negative feedback ( nadir LH as % of baseline LH); Test type: Superiority or Other; p = 0.90, ANOVA
Statistical Analysis 2: Comparison: Younger PMW vs Older PMW; positive feedback; Test type: Superiority; p < 0.03, ANOVA — a priori threshold for significance is p<0.05

2. Primary Outcome: Effect of Aging on Estrogen Positive Feedback on LH
Description: LH area under the curve in response to estrogen positive feedback. Area under the curve was calculated from blood samples drawn every 4 hours from the onset of positive feedback until the end of the study (120 min). The onset of positive feedback is defined as the time when LH first exceeds mean + 2SD of the previous three time points and shows a sustained rise.
Time Frame: Onset of surge (average of 61 hr from beginnning of infusion until the end of the study (120 hr)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: IU*hr/L
Arm/Group | Young Postmenopausal Women | Older Postmenopausal Women
Number analyzed (Participants) | 11 | 9
IU*hr/L | 4544.6 (636.3) | 2885.5 (316.7)
Statistical Analysis 1: Comparison: Young Postmenopausal Women vs Older Postmenopausal Women; Test type: Superiority; p = 0.03, ANOVA — a priori significance level p<0.05

3. Secondary Outcome: 18 FDG Uptake at the Pituitary During Estrogen Infusion: LH Negative Feedback
Description: Regional cerebral glucose metabolism (rCMRglu) is used as a measure of neuronal metabolic activity and calculated as average uptake (voxels) of 18 flurodeoxyglucose within the region of interest (ROI) and expressed simply as units. Normalized uptake refers to co-registration of the PET with the MRI to provide more accurate anatomic correlates.
Time Frame: Baseline vs 24 hr after the onset of steroid infusion
Population: postmenopausal women
Measure: Mean (Standard Error); unit: units
Groups:
- Baseline Pituitary: 18 FDG uptake at the pituitary at baseline
- Negative Feedback Pituitary: 18 FDG uptake at the pituitary at 24 hr associated with estrogen induced negative feedback on LH
Arm/Group | Baseline Pituitary | Negative Feedback Pituitary
Number analyzed (Participants) | 11 | 11
units | 45.8 (4.5) | 48.4 (4.0)
Statistical Analysis 1: Comparison: Baseline Pituitary vs Negative Feedback Pituitary; Test type: Superiority; p = 0.49, t-test, 2 sided — threshold for significance p<0.05

4. Secondary Outcome: 18 FDG Uptake at the Hypothalamus During Estrogen Infusion: LH Negative Feedback
Description: as for outcome 3
Time Frame: 0 vs 24 hr
Population: postmenopausal women
Measure: Mean (Standard Error); unit: units
Groups:
- Baseline Hypothalamus: 18 FDG uptake at the hypothalamus at baseline
- Negative Feedback Hypothalamus: 18 FDG uptake at the at the hypothalamus at 24 hr associated with estrogen induced negative feedback on LH
Arm/Group | Baseline Hypothalamus | Negative Feedback Hypothalamus
Number analyzed (Participants) | 11 | 11
units | 69.0 (3.3) | 63.1 (2.8)
Statistical Analysis 1: Comparison: Baseline Hypothalamus vs Negative Feedback Hypothalamus; Test type: Superiority; p < 0.02, t-test, 2 sided — a priori threshold for significance p<0.05

5. Secondary Outcome: 18 FDG Uptake at the Pituitary During Estrogen Infusion: LH Positive Feedback
Description: as for outcome 3
Time Frame: 24 hr vs 72 hr
Population: postmenopausal women
Measure: Mean (Standard Error); unit: units
Groups:
- Pituitary at 24 hr: 18 FDG uptake at the pituitary at 24 hr
- Pituitary at 72 hr: 18 FDG uptake at the pituitary at 72 hr associated with estrogen induced positive feedback on LH
Arm/Group | Pituitary at 24 hr | Pituitary at 72 hr
Number analyzed (Participants) | 11 | 11
units | 48.0 (4.0) | 54.3 (4.4)
Statistical Analysis 1: Comparison: Pituitary at 24 hr vs Pituitary at 72 hr; Test type: Superiority; p < 0.03, t-test, 2 sided

6. Secondary Outcome: 18 FDG Uptake at the Hypothalamus During Estrogen Infusion: LH Positive Feedback
Description: as for outcome 3
Time Frame: 24 vs 72 hr
Population: postmenopausal women
Measure: Mean (Standard Error); unit: unit
Groups:
- Hypothalamus at 24 hr: 18 FDG uptake at the hypothalamus at 24 hr
- Hypothalamus 72 hr: 18 FDG uptake at the pituitary at 72 hr associated with estrogen induced positive feedback on LH
Arm/Group | Hypothalamus at 24 hr | Hypothalamus 72 hr
Number analyzed (Participants) | 11 | 11
unit | 63.1 (2.8) | 66.2 (3.7)
Statistical Analysis 1: Comparison: Hypothalamus at 24 hr vs Hypothalamus 72 hr; Test type: Superiority; p = 0.07, t-test, 2 sided — a priori significance set at p<0.05

ADVERSE EVENTS:
Time Frame: 60 days for each subject; 4 years in total
Description: As in clinicaltrials.gov
Arm/Group | Younger PMW | Older PMW
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 2/13 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Younger PMW (N=13) | Older PMW (N=12)
anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — decrease in hemoglobin below pre-specified level
vasomotor symptoms (Vascular disorders) | 2 (2) | 0 (0) — mild vasomotor symptoms during estradiol infusion

LIMITATIONS AND CAVEATS:
PET scan data addresses hypothalamic vs pituitary sites of negative and positive estrogen feedback on LH, but there was insufficient power to address the effect of aging on these secondary measures..

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No